CLINICAL TRIAL: NCT06749587
Title: A Prospective, Multi-center, Randomized, No-Treatment Controlled, Evaluator-Blinded, Superiority Clinical Investigation of the Safety and Effectiveness of TEOSYAL RHA® 1 for the Correction of Moderate to Severe Tissue Volume Deficiency in the Infraorbital Region in Chinese Adults
Brief Title: TEOSYAL RHA® 1 for the Correction of Moderate to Severe Tissue Volume Deficiency in the Infraorbital Region in Chinese Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Teoxane SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TEO-TPRL-2401
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Infraorbital Hollows
Keywords: Dermal Filler; Hyaluronic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinded-Live Evaluator (BLE)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEOSYAL RHA® 1 (Experimental)
  Interventions: Device: TEOSYAL RHA® 1
- Control group (non treated) (No Intervention)

INTERVENTIONS:
Device: TEOSYAL RHA® 1 — Product injection in infraorbital hollows
  TEOSYAL RHA® 1 is a sterile, transparent, non-pyrogenic, viscoelastic gel made of Hyaluronic Acid (HA) of non-animal origin
  Arms: TEOSYAL RHA® 1

SUMMARY:
This is a prospective, multi-center, randomized, no-treatment controlled, evaluator-blinded clinical investigation to identify whether TEOSYAL RHA® 1 is superior to no treatment for the correction of moderate to severe tissue volume deficiencies in the infraorbital region in Chinese adults.

Eligible subjects will be enrolled and randomized either to the treatment group or control group in a 3:1 ratio on Day 0. Each subject assigned to the treatment group will receive TEOSYAL RHA® 1 in both Infraorbital Hollows (IOH), whereas subjects assigned to the control group will not receive any treatment.

The subjects in the treatment group will be treated with RHA1 for the treatment of moderate to severe tissue volume deficiencies in the infraorbital region on Day 0.

All treated subjects will return to the site at 2, 4, 12, 24, 36, and 52 weeks after the last treatment for effectiveness and safety assessments. Each treated subjects will receive a safety phone call 3 days after the initial treatment at baseline, and after the touch-up treatment, if any. Their participation in the trial ends after the completion of the follow up period.

All non treated subjects (control group) will return to the site at 2, 4, and 12 weeks after randomization for effectiveness and safety assessments. Their participation in the investigation ends after the effectiveness and safety assessments at 12 weeks after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese male and female, 18 years of age or older.
2. Subject seeking treatment of moderate to severe tissue volume deficiencies in the infraorbital region.
3. Subjects with a grade of 2 (moderate) or 3 (severe) on the TIOHS for both eyes, as determined on assessments by the Treating Investigator (TI) and BLE.
4. Subject willing to abstain from all other facial aesthetic procedures/therapies that could interfere with effectiveness evaluations (e.g., dermal fillers outside of this investigation, toxin treatments, facial ablative or fractional laser, Intense Pulsed Light [IPL], microdermabrasion, chemical peels, skin bleaching agents, non-ablative laser, or energy-based device for skin-tightening, surgical procedures, etc.) during participation in the investigation.
5. Woman of childbearing potential agree to use contraception during the investigation.
6. Subject understands and is able to follow instructions and complete all scheduled visits.
7. Subjects who voluntarily decided to participate in the investigation and signed the informed consent.

Exclusion Criteria:

1. Known hypersensitivity or previous allergic reaction to any component of the study device.
2. Known sensitivity to local anesthetics of the amide type, history of multiple severe allergies, or history of anaphylactic shock.
3. History of active chronic debilitating systemic disease that, in the opinion of the investigator, would make the subject a poor candidate in the study.
4. History of connective tissue disease.
5. Clinically significant alcohol or drug abuse, or history of poor cooperation or unreliability.
6. Subjects who participated in other clinical investigation within 30 days, or in an exclusion period from a previous study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-03-12 (Estimated); Study Completion 2026-01-12 (Estimated)

PRIMARY OUTCOMES:
TIOHS = Teoxane Infraorbital Hollows Scale (grade 0 = no visible infraorbital hollow ; grade 4 = very severe infraorbital hollow) | 12 weeks after the last treatment for the treatment group / 12 weeks after randomization for the control group
  Proportion of responders, defined by at least 1-grade improvement in both eyes from baseline 5-point TIOHS, as assessed by the BLE at 12 weeks after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Second Provincial General Hospital, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No